CLINICAL TRIAL: NCT01360359
Title: Recurrent Low Back Pain: Linking Mechanism to Outcomes (RCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sheri Silfies, Principal Investigator, Drexel University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: K01HD053632 (NIH); K01HD053632 (NIH)
Record Dates: First submitted 2011-05-24; First posted 2011-05-25 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Low Back Pain
Keywords: low back pain; core stabilization; trunk muscle exercises; physical therapy; RCT
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Core Stabilization (Experimental): 8-week core stabilization program in 3 stage that emphasizes use of specific local trunk stabilizing muscles to restore active control and stability to the trunk.
  8-week exercise program, 1-2 sessions/ week, 30-60 minute sessions
  Interventions: Other: Core Stabilization
- Trunk Motion and Fitness (Active Comparator): 8-week exercise program in 3 stages emphasizing spine motion, general trunk flexibility and strengthening and cardiovascular fitness.
  8-week exercise program, 1-2 sessions/ week, 30-60 minute sessions
  Interventions: Other: Trunk Motion and Fitness

INTERVENTIONS:
Other: Core Stabilization — 3 Stages: Stage 1: emphasis on neutral spine position, co-contraction of stabilizing muscles with performance feedback through observation and palpation for correct muscle activation; patient education
  Stage 2: promotes maintenance of co-contraction while performing movements of the arms/legs and trunk progressing to preformance of these exercises on unstable surfaces; trunk muscle conditioning also emphasized; feedback gradually reduced.
  Stage 3: emphasis on maintenance of co-contraction while performing functional activities; stable and unstable surfaces; use of perturbation and random practice to enhance motor learning.
  Arms: Core Stabilization
Other: Trunk Motion and Fitness — 3 Stages: Stage 1: reducing pain and restoring spine motion and flexibility; patient education
  Stage 2: trunk muscle conditioning exercises
  Stage 3: trunk muscle conditioning and cardiovascular conditioning exercises
  Arms: Trunk Motion and Fitness

SUMMARY:
The purpose of this randomized clinical trial of low back pain exercise programs is to determine if trunk control can be changed by core stabilization exercises. The proposed mechanism of pain reduction and functional improvement of core stabilization exercises is that it enhances trunk movement and muscle control. This study will provide preliminary evidence of the link between patient outcomes and treatment mechanisms.

The investigators hypothesize that:

* both treatment groups will demonstrate significant improvements in pain and function;
* only subjects in the core stabilization group will demonstrate significant improvements in trunk movement and muscle control.

ELIGIBILITY:
Inclusion Criteria:

1. duration of the current episode less than 3 months,
2. average pain intensity over past 2 weeks greater than 4 on an 11 point (0 = no pain, 10 = worst pain ever) verbal pain rating scale,
3. self-report global function less than 80% (0-100 %, 100% = normal pain free function)
4. Oswestry Index > 19%
5. no physical therapy or chiropractic treatment for the current episode of low back pain.
6. clinical diagnosis of poor trunk control/ clinical lumbar instability needs to be met based upon completion of specific physical therapy examination finding

Exclusion Criteria:

1. permanent structural spinal deformity (e.g., scoliosis),
2. spinal fracture or history of spinal fracture,
3. osteoporosis,
4. inflammatory joint disease,
5. signs of systemic illness or suspected non-mechanical LBP (spinal tumor or infection),
6. previous spinal surgery,
7. frank neurological loss, i.e., weakness and sensory loss in a NR distribution,
8. pain or paresthesia below the knee,
9. leg length discrepancy of greater than 2.5 cm,
10. history of neurologic disease that required hospitalization,
11. active treatment of another medical illness that would preclude participation in any aspect of the study,
12. pregnancy,
13. vestibular dysfunction,
14. extreme psychosocial involvement
15. allergies to medical tape or adhesives
16. Body mass index greater than 30 kg/m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Trunk Neuromuscular Control | Baseline, 8 weeks
  Using surface EMG, kinematics and force parameters. Trunk neuromuscular control is characterized and compared between groups and pre/post intervention.

SECONDARY OUTCOMES:
Clinical Outcomes | Baseline, 8-weeks
  Oswestry Disability Index- measure of self-perceived functional limitations NPRS- numeric pain index

CONTACTS AND LOCATIONS:
Overall Officials: Sheri P. Silfies, PT, PhD, Principal Investigator — Drexel University
Locations (2):
- United States (2):
  - Drexel University Physical Therapy, Philadelphia, Pennsylvania
  - Optimum Physical Therapy Associates, West Chester, Pennsylvania